CLINICAL TRIAL: NCT02636647
Title: Safety and Tolerability of Fecal Microbiota Transplantation in Cirrhosis and Hepatic Encephalopathy
Brief Title: Fecal Transplant in Recurrent Hepatic Encephalopathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jasmohan Bajaj (U.S. Federal Agency)
Collaborators: OpenBiome (Industry)
Responsible Party: Sponsor-Investigator, Jasmohan Bajaj, MD, Hunter Holmes Mcguire Veteran Affairs Medical Center
Organization: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BAJAJ0021
Record Dates: First submitted 2015-12-16; First posted 2015-12-22 (Estimated); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Hepatic Encephalopathy; Cirrhosis
Keywords: hepatic encephalopathy; fecal transplant; cirrhosis
MeSH Terms: conditions — Hepatic Encephalopathy; Fibrosis | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FMT (Active Comparator): Fecal transplant via enema once
  Interventions: Biological: Fecal transplant
- No treatment (No Intervention): No transplant performed

INTERVENTIONS:
Biological: Fecal transplant
  Arms: FMT

SUMMARY:
Randomized, open-label safety, tolerability study with exploratory endpoints and pathophysiological evaluation of the FMT

Two groups of outpatients with cirrhosis will be randomized using random sequence generator into no-treatment and FMT groups.

DETAILED DESCRIPTION:
Group 1 (FMT group) will undergo the following procedures

Pre-FMT preparation:

We will obtain written informed consent per the IRB guidelines. After the patients are consented and are eligible, we will perform a detailed medical history and physical exam at day 0. We will also perform cognitive testing. As in prior studies, we will prescribe patients an antibiotic regimen. Drawing from ecological principles of microbial niche environments and data from recurrent Clostridium difficile infection, pre-treatment antibiotics are likely to increase the probability of disrupting the hosts intrinsic microbiota and creating an opportunity for a 'healthy' microbiota from the FMT to engraft.

After antibiotics and on the day of FMT:

At day 5, we will re-evaluate patients with a directed interval history and focused physical exam as needed. After ensuring that they are still candidates according to the inclusion/exclusion criteria, we will collect stool, urine and blood again for pre-FMT evaluation and urine for pregnancy tests from eligible women. Cognitive testing will be performed again.

Preparation and handling of stool for FMT infusion

Standard protocol for handling bio-hazardous material will be employed in order to avoid contamination and risk to healthcare handlers. Sterile microbiological technique will be employed during material transfer peri-procedure.

At that point we will provide the fecal material using universal precautions to a standard retention enema bag. The procedure will be completed by a trained Registered Nurse, Nurse practitioner, or physician in an outpatient clinic, endoscopy recovery area, or standard endoscopy unit.

The following will be recorded in all FMTs

* Dose
* Unit ID/Lot# of each treatment
* Expiration Date
* Storage Condition
* FMT retention time (in minutes)

Number of FMT: One administration Duration of Follow-up after FMT: 5 months

Follow-up after FMT:

We will see the patient in clinic the day following FMT (day 6 or FMT+1), day 12 (FMT+7), day 20 (FMT+15), and day 35 (FMT+30), at which point a detailed history regarding abdominal symptoms, evaluation of infectious complications, hospitalizations or complications of cirrhosis.

Visits on day 6, day 12 and day 35 will be purely safety associated while, on the day 20 visit, we will repeat the pathophysiological studies.

In order to ensure that we have enough samples, in case patients are not able to return at day 20, we will also collect all samples at day 12, but will only analyze them in case the day 20 visit does not occur.

These visits, apart from the visit after FMT, will be ±2 days for patient convenience.

At 5 months post-FMT, subjects will be followed up with a phone call to evaluate potential SAEs, new onset of transmitted infections, new onset or significant worsening of chronic medical conditions or suspected unexpected serious adverse reactions that have occurred in between 35 days and 5 months for reporting purposes.

Samples collected at baseline (before FMT), after antibiotics and at day 15 will be:

1. Stool
2. Blood
3. Urine

Group 2: No treatment arm The group 2 will undergo all sample collections, follow-up and cognitive testing as in group 1 but without the 5-day antibiotic therapy or the FMT. In addition, we will also not perform the sample collection that is done after 5 days of antibiotics in this group since no reasonable change in microbiota are expected over 5 days without antibiotics. The follow-up of this group will be same as that of the FMT group.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis diagnosed by either of the following in a patient with chronic liver disease

  * Liver Biopsy
  * Radiologic evidence of varices, cirrhosis or portal hypertension
  * Laboratory evidence of platelet count <100,000 or AST/ALT ratio>1
  * Endoscopic evidence of varices or portal gastropathy
* At least two episodes of hepatic encephalopathy, one within the last year but not within the last month (patient can be on lactulose and rifaximin)
* Age between 21 and 75
* Able to give written, informed consent (demonstrated by mini-mental status exam>25 at the time of consenting)

Exclusion Criteria:

* MELD score >17
* WBC count <1000 cells/mm3
* Platelet count<50,000/mm3
* On the liver transplant list
* TIPS in place
* No HE episode within a month prior to the study
* Patients allergic to ciprofloxacin, penicillins or metronidazole
* Currently on absorbable antibiotics
* Infection at the time of the FMT (diagnosed by blood culture positivity, urinalysis, paracentesis as needed)
* Hospitalization for any non-elective cause within the last 3 months
* Patients who are aged >75 years
* Patients who are pregnant or nursing (will be checked using a urine pregnancy test)
* Patients who are incarcerated
* Patients who are incapable of giving their own informed consent
* Patients who are immuno-compromised due to the following reasons:

  * HIV infection (any CD4 count)
  * Inherited/primary immune disorders
  * Current or recent (<3 mos) treatment with anti-neoplastic agent
  * Current or recent (<3 mos) treatment with any immunosuppressant medications [including but not limited to monoclonal antibodies to B and T cells, anti-TNF agents, glucocorticoids, antimetabolites (azathioprine, 6-mercaptopurine), calcineurin inhibitors (tacrolimus, cyclosporine), mycophenolate mofetil]. Subjects who are otherwise immunocompetent and have discontinued any immunosuppressant medications 3 or more months prior to enrollment may be eligible to enroll.
* Patients with a history of severe (anaphylactic) food allergy
* Patients who have previously undergone FMT
* Patients on renal replacement therapy
* Patients who are unwilling or unable to hold the enemas
* Patients with untreated, in-situ colorectal cancer
* Patients with a history of chronic intrinsic GI diseases such as inflammatory bowel disease (ulcerative colitis, Crohn's disease or microscopic colitis) , eosinophilic gastroenteritis, celiac disease or irritable bowel syndrome
* Major gastro-intestinal or intra-abdominal surgery in the last three months
* Unable to comply with protocol requirements
* Patients who are American Society of Anesthesiologists (ASA) Physical Status classification IV and V
* Patients with acute illness or fever on the day of planned FMT will be excluded with the option of including that subject at a future date
* Any conditions for which, in opinion of MD, the treatment may pose a health risk
* C. difficile in the stool at baseline (qPCR)
* Grade 2-4 or complicated hemorrhoids

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | 5 months
  Defined by the rate of development of FMT-related SAE and withdrawal from the study in cirrhotic subjects

SECONDARY OUTCOMES:
Microbiota composition and function | 15 days
  Deep sequencing of the microbiota and urinary metabolomics at baseline and post-FMT
Cognitive functioning | 15 days
  Computerized and paper-pencil test battery

CONTACTS AND LOCATIONS:
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No